CLINICAL TRIAL: NCT05259696
Title: A Phase 1/2, Open-Label, Single-Arm, Dose-Escalation and Dose-Expansion Study of the Safety, Tolerability, Pharmacokinetic, and Antitumor Activity of E-602 as a Single Agent and in Combination With Cemiplimab in Patients With Advanced Cancers
Brief Title: Glycan Mediated Immune Regulation With a Bi-Sialidase Fusion Protein (GLIMMER-01)
Acronym: GLIMMER-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Palleon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PAL-E602-001
Record Dates: First submitted 2022-02-11; First posted 2022-02-28 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Oncology; Melanoma; Ovarian Cancer; NSCLC; Non Small Cell Lung Cancer; Colorectal Cancer; Pancreatic Cancer; Cancer; CRC; Colon Cancer; Breast Cancer; Gastric Cancer; EGJ; Esophagogastric Junction Cancer; Head and Neck Cancer; Urothelial Cancer; Bladder Cancer
Keywords: Cancer; Bi-Sialidase; Anti-Tumor; E-602; Cemiplimab
MeSH Terms: conditions — Neoplasms; Melanoma; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Urinary Bladder Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: Phase 1: The study uses a modified 3+3 design with 5 planned dose levels of E-602 as monotherapy and 2 planned dose levels of E-602 in combination with cemiplimab. Phase 2: Consists of dose-expansion and will use the recommended Phase 2 dose level for E-602 as monotherapy and in combination with cemiplimab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation - Monotherapy (Experimental): Subjects will receive E-602 as monotherapy.
  Planned monotherapy dose levels: 1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg, and 30 mg/kg.
  Interventions: Biological: E-602
- Dose Escalation - Combination (Experimental): Subjects will receive E-602 in combination with cemiplimab.
  E-602 dose(s): Will be initiated at dose level(s) that have previously completed dosing and DLT assessments as monotherapy.
  Cemiplimab dose: 350 mg.
  Interventions: Biological: E-602; Biological: Cemiplimab
- Expansion - Monotherapy (Experimental): Subjects will receive E-602 as monotherapy at the recommended Phase 2 dose determined in Phase 1.
  Interventions: Biological: E-602
- Expansion - Combination (Experimental): Subjects will receive E-602 in combination with cemiplimab.
  E-602 dose: Subjects will receive E-602 at the recommended Phase 2 dose determined in Phase 1 in combination with cemiplimab.
  Cemiplimab dose: 350 mg.
  Interventions: Biological: E-602; Biological: Cemiplimab

INTERVENTIONS:
Biological: E-602 — Subjects will receive E-602 (administered weekly, via IV infusion).
Biological: Cemiplimab — Subjects will receive cemiplimab (administered once every 3 weeks, via IV infusion).
  Other Names: Libtayo; REGN2810
  Arms: Dose Escalation - Combination; Expansion - Combination

SUMMARY:
This is a Phase 1/2, first-in-human, open-label, dose escalation and dose-expansion study of E-602, administered alone and in combination with cemiplimab.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the safety, tolerability, PK, pharmacodynamics, and antitumor activity of E-602 in subjects with advanced cancers.

Phase 1 of the study consists of dose escalation cohorts of E-602 as a monotherapy and in combination with cemiplimab. Dose escalation will utilize a modified 3+3 design. Any Phase 1 cohort may be backfilled, up to a total of 15 subjects to obtain additional safety, PK, and pharmacodynamic data at a particular dose level. Phase 1 will treat subjects with melanoma, ovarian cancer, non-small cell lung cancer (NSCLC), colorectal cancer, pancreatic cancer, breast cancer, gastric/esophagogastric junction (EGJ) cancer, head and neck cancer, or urothelial cancer. The safety and pharmacodynamic data will be evaluated to identify the maximum tolerated dose and recommended Phase 2 dose level for E-602 as monotherapy and in combination with cemiplimab.

Phase 2 consists of dose-expansion disease cohorts in subjects with 3 types of advanced tumors: melanoma, NSCLC, and a third type to be determined (ovarian, colorectal, pancreatic, breast, gastric/EGJ, head and neck, or urothelial) based on available data. Phase 2 includes cohorts of E-602 as monotherapy and E-602 in combination with cemiplimab. For each cohort in Phase 2, Simon's minimax 2-stage design will be used.

The study is seeking to enroll a total of up to 273 subjects (up to 87 in Phase 1 and up to 186 in Phase 2). Subjects will participate in the study for about 16 months.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects with advanced or relapsed/refractory melanoma, ovarian cancer, NSCLC, colorectal cancer, pancreatic cancer, breast cancer, gastric/esophagogastric junction (EGJ) cancer, head and neck cancer, or urothelial cancer who have failed prior therapies.

   a. Subjects with melanoma, NSCLC, head and neck cancer, urothelial cancer, or mMSI-H or dMMR colorectal cancer must have had prior anti-PD-(L)1 pathway therapy and been deemed resistant (had progression on therapy or within 3 months of discontinuation of therapy).
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Subject has disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
4. Adequate bone marrow, coagulation, renal function, and liver function as determined by laboratory tests

Key Exclusion Criteria:

1. For cohorts receiving E-602 and cemiplimab combination therapy:

   1. Prior moderate or severe hypersensitivity to cemiplimab or its formulation
   2. History of severe (≥ Grade 3) autoimmune complications or discontinuation due to toxicity following treatment with an anti-PD-(L)1 pathway therapy as a monotherapy, with the exception of asymptomatic Grade 3 elevations in lipase and/or amylase not associated with clinical manifestations of pancreatitis.
   3. Subject has an active autoimmune disease. The following are not exclusionary: vitiligo, type 1 diabetes, autoimmune endocrinopathies that are stable on hormone replacement therapy, or psoriasis that does not require systemic treatment.
   4. Previously received idelalisib.
2. History of age-related macular degeneration (AMD).
3. Recent surgery, treatment with another investigational agent, active infection, non-healing wound or uncontrolled bleeding/bleeding diathesis.
4. Received a vaccine or prior radiotherapy within 14 days prior to Cycle 1 Day 1.
5. Prior history of interstitial lung disease that required steroids or ≥ Grade 2 immune-related pneumonitis or has current non-infectious pneumonitis or interstitial lung disease. Subject has a history of ≥Grade 3 radiation pneumonitis, or Grade 2 radiation pneumonitis that has been active within the last 6 months.
6. Untreated brain metastases.
7. A known primary malignancy that is progressing or has required active treatment within the past 3 years.
8. Subject is taking the equivalent of >10 mg/day oral prednisone or on systemic immunosuppressive therapy.
9. Subject has had an allogeneic tissue or organ transplantation.
10. History of thromboembolic event unless the event occurred > 6 months from Cycle 1 Day 1 and the subject is on anti-coagulation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Stanford Health Care, Stanford, California
  - Yale University Cancer Center, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Columbia University, New York, New York
  - Providence Cancer Institute, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- E-602 1 mg/kg: Participants received 1 mg/kg E-602 monotherapy administered weekly via IV infusion.
- E-602 3 mg/kg: Participants received 3 mg/kg E-602 monotherapy administered weekly via IV infusion.
- E-602 10 mg/kg: Participants received 10 mg/kg E-602 monotherapy administered weekly via IV infusion.
- E-602 20 mg/kg: Participants received 20 mg/kg E-602 monotherapy administered weekly via IV infusion.
- E-602 30 mg/kg: Participants received 30 mg/kg E-602 monotherapy administered weekly via IV infusion.
- E-602 20 mg/kg in Combination With Cemiplimab: Participants received 20 mg/kg E-602 monotherapy administered weekly via IV infusion. They also received 350 mg cemiplimab administered every 3 weeks via IV infusion.
Period: Overall Study
Arm/Group | E-602 1 mg/kg | E-602 3 mg/kg | E-602 10 mg/kg | E-602 20 mg/kg | E-602 30 mg/kg | E-602 20 mg/kg in Combination With Cemiplimab
Started | 5 | 4 | 9 | 15 | 15 | 21
Completed | 5 | 4 | 9 | 15 | 15 | 21
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was used for analysis purposes.
Groups:
- Total: Total of all reporting groups
Arm/Group | E-602 1 mg/kg | E-602 3 mg/kg | E-602 10 mg/kg | E-602 20 mg/kg | E-602 30 mg/kg | E-602 20 mg/kg in Combination With Cemiplimab | Total
Number analyzed (Participants) | 5 | 4 | 9 | 15 | 15 | 21 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (10.79) | 60.0 (11.17) | 57.9 (12.39) | 59.1 (9.36) | 62.1 (10.25) | 66.5 (10.31) | 61.7 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 7 | 7 | 11 | 36
  Male | 3 | 0 | 4 | 8 | 8 | 10 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 2 | 2 | 1 | 5
  Black or African American | 0 | 0 | 1 | 1 | 0 | 1 | 3
  White | 3 | 4 | 7 | 11 | 13 | 18 | 56
  Other | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Not Reported | 1 | 0 | 1 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced AEs or SAEs
Description: Number of participants who experienced an adverse events (AEs) or a serious adverse event (SAE)
Time Frame: 15 Months
Measure: Count of Participants; unit: Participants
Arm/Group | E-602 1 mg/kg | E-602 3 mg/kg | E-602 10 mg/kg | E-602 20 mg/kg | E-602 30 mg/kg | E-602 20 mg/kg in Combination With Cemiplimab
Number analyzed (Participants) | 5 | 4 | 9 | 15 | 15 | 21
Participants
  Participants with any Treatment Emergent AE | 5 | 4 | 8 | 15 | 15 | 20
  Participants with any Serious AE | 3 | 1 | 1 | 6 | 5 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the treatment period, up to 12 months, and up to 3 months after treatment discontinuation.
Description: Adverse Events were graded using CTCAE v5.0
Arm/Group | E-602 1 mg/kg | E-602 3 mg/kg | E-602 10 mg/kg | E-602 20 mg/kg | E-602 30 mg/kg | E-602 20 mg/kg in Combination With Cemiplimab
All-Cause Mortality (participants affected / at risk) | 5/5 | 1/4 | 7/9 | 9/15 | 6/15 | 5/21
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/4 | 1/9 | 6/15 | 5/15 | 5/21
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 8/9 | 15/15 | 15/15 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-602 1 mg/kg (N=5) | E-602 3 mg/kg (N=4) | E-602 10 mg/kg (N=9) | E-602 20 mg/kg (N=15) | E-602 30 mg/kg (N=15) | E-602 20 mg/kg in Combination With Cemiplimab (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-602 1 mg/kg (N=5) | E-602 3 mg/kg (N=4) | E-602 10 mg/kg (N=9) | E-602 20 mg/kg (N=15) | E-602 30 mg/kg (N=15) | E-602 20 mg/kg in Combination With Cemiplimab (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 6 | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 4 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 1 | 4
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 4
Fatigue (General disorders) | 1 | 1 | 3 | 3 | 4 | 7
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 10 | 10 | 9
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 3 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 3 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 4 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 2 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 3 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT05259696/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT05259696/SAP_001.pdf